CLINICAL TRIAL: NCT01776346
Title: Barrett's Esophagus Patient Registry
Acronym: BPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Chin Hur, Principal Investigator; MD, MPH, Massachusetts General Hospital
Other Study IDs: 2010P002224
Record Dates: First submitted 2013-01-22; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma; Gastroesophageal Reflux
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Serum (from whole blood), plasma (from whole blood), tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Barrett's Esophagus/Esophageal Adenocarcinoma: Patients who have Barrett's esophagus or esophageal adenocarcinoma.
- Healthy control

SUMMARY:
The ultimate goal of the Barrett's Esophagus Patient Registry is to help develop more effective targeted screening strategies and treatment options for Barrett's esophagus and esophageal adenocarcinoma (EAC). We plan to do by developing a registry that will serve as a platform. Examples of analyses could include identifying genetic determinants and biomarkers that predict BE, progression of BE to EAC, as well as the response to therapies.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's (BE): Patients who have Barrett's esophagus (all stages: Barrett's metaplasia, low-grade dysplasia, high-grade dysplasia) based upon standard endoscopic and histologic criteria.
* Adenocarcinoma (EAC): Patients who have esophageal adenocarcinoma.
* The control cohort will include patients ages 18 and older with no prior history of BE and EAC. These may include patients who are being seen or have been previously seen at MGH GI Associates for conditions including gastroesophageal reflux disease, peptic esophagitis, eosinophilic esophagitis, esophageal motility disorders such as achalasia and nutcracker esophagus.

Exclusion Criteria:

* Inability or unwillingness to provide blood samples.
* History of known bleeding disorders.
* Currently awaiting organ transplantation.
* Having an acute or severe chronic illness such as congestive heart failure or any other condition that would prohibit performing the endoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been seen at Massachusetts General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2011-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression to esophageal adenocarcinoma | 5 years (on average although follow-up will continue)

SECONDARY OUTCOMES:
Identify and validate genetic determinants that predict progression of BE to EAC and predict response to BE therapy | 5 years on average
Evaluate the natural history of BE with and without treatment based on clinical, functional and economic outcomes of the cases | 5 years on average

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States